CLINICAL TRIAL: NCT00005386
Title: Biobehavioral Determinants of Obesity in Black Women
Status: Completed | Type: Observational
Sponsor: University of Memphis (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4292; R01HL053261 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2004-08

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Obesity; Telangiectasis
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Obesity; Telangiectasis

SUMMARY:
To examine the biobehavioral determinants of obesity in Black as compared with white women.

DETAILED DESCRIPTION:
BACKGROUND:

Behavioral medicine surveys consistently find that obesity is a treatment-resistant disease that continues to be a significant health problem and that the incidence of obesity is much higher in Blacks relative to whites in general, and even higher in Black women relative to white women. In fact, an NIH Program Announcement (PA-91-99), stated that "Obesity in adults has not declined in the past three decades" and "Obesity is particularly prevalent in minority populations, especially among minority women." Obesity is an independent risk factor for cardiovascular disease, stroke, and hypertension. Obesity is a complex phenomenon involving behavioral, lifestyle, and complex biobehavioral mechanisms. In 1995, there were no prospective studies that simultaneously evaluated a systematic set of psychosocial variables with energy balance (dietary intake, physical activity, resting metabolic rate) determinants that may account for the increased risk for obesity in African-American versus Euro-American women.

DESIGN NARRATIVE:

After subjects were recruited, psychosocial and energy balance (dietary intake, physical activity, metabolic rate) baseline measures were related to levels of body fat as measured by DEXA (dual electron X-ray absorptiometry). The role of these variables were evaluated prospectively to adiposity changes in both white and Black women over a 24-month period.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1995-09; Study Completion 1998-08

CONTACTS AND LOCATIONS:
Overall Officials: Robert Klesges — University of Memphis

REFERENCES:
- [Background] Scarinci IC, Slawson DL, Watson JM, Klesges RC, Murray DM. Socioeconomic status, ethnicity, and health care access among young and healthy women. Ethn Dis. 2001 Winter;11(1):60-71. PMID 11289253
- [Background] Scarinci IC, Watson JM, Slawson DL, Klesges RC, Murray DM, Eck-Clemens LH. Socioeconomic status, ethnicity, and environmental tobacco exposure among non-smoking females. Nicotine Tob Res. 2000 Nov;2(4):355-61. doi: 10.1080/713688150. PMID 11197316